CLINICAL TRIAL: NCT03727724
Title: Phase II Single Arm Study of Afatinib in Combination With Cetuximab in EGFR Exon 20 Insertion Positive Non-small-cell Lung Cancer
Brief Title: Afatinib and Cetuximab in Epidermal Growth Factor Receptor (EGFR) Exon 20 Insertion Positive Non-small-cell Lung Cancer
Acronym: AFACET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Boehringer Ingelheim (Industry); Merck Serono International SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M18ACX
Record Dates: First submitted 2018-09-03; First posted 2018-11-01 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Afatinib plus cetuximab (Experimental): Afatinib, 40 mg once daily, orally.
  Cetuximab, 500 mg/m² intravenously, every 2 weeks.
  Treatment will be continued until tumor progression (according RECIST v1.1) confirmed by tumor imaging, unacceptable toxicity, or death occurs.
  Interventions: Drug: Afatinib; Drug: Cetuximab

INTERVENTIONS:
Drug: Afatinib — Tablet
Drug: Cetuximab — Injection

SUMMARY:
This is a single arm open-label multi-center phase II study, investigating disease control rate after 18 weeks of treatment with afatinib/cetuximab combination therapy in patients with advanced non-small cell lung cancer (NSCLC) harboring an EGFR exon 20 insertion.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically confirmed stage IV non-small cell lung cancer, harboring an EGFR exon 20 insertion mutation.
* 18 years or older at time of study entry.
* Life expectancy of at least three months.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 (see Appendix 1).
* Measurable disease, according to RECIST 1.1.
* At baseline adequate fresh or archived tissue from a histological biopsy or a cellblock obtained by fine needle aspiration of a tumor lesion that is not radiated prior to biopsy, must be available. Baseline tissue samples must have been obtained after the last line of systemic therapy prior to study entry.
* Adequate normal organ and marrow function as defined below:
* Absolute leukocyte count ≥ 3 x 109/L (> 3000 per mm3)
* Platelet count ≥ 75 x 109/L (>75,000 per mm3)
* Aspartate amino transferase (AST) or alanine amino transferase (ALT) ≤ 3 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x upper limit of normal (ULN).
* Serum creatinine clearance >30 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance.
* Women of child-bearing potential: these subjects must have a negative serum pregnancy test within 7 days prior to the first dose of study treatment and agree to use highly effective contraception, as defined in section 5.2.2, from 7 days prior to enrollment, throughout the treatment period and for seven months after completion of the treatment with cetuximab.
* Males must agree to take appropriate precautions to avoid fathering a child from the first dose of study treatment through 3 months after the final administration of investigational drugs.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Ability to give written informed consent before patient registration.

Exclusion Criteria:

* Participation in another clinical study with an investigational product during the last 2 weeks.
* Prior treatment with EGFR targeting antibodies (prior treatment with EGFR TKI's is allowed).
* Other active malignancy.
* History of hypersensitivity to afatinib or cetuximab.
* Major surgery (excluding diagnostic procedures e.g. mediastinoscopy or video assisted thoracic surgery (VATS) biopsy) within 28 days of the start of study treatment.
* Radiotherapy less than two weeks prior to the start of study treatment.
* Symptomatic brain metastases.
* Breast feeding is not allowed during study treatment.
* Uncontrolled intercurrent illness including ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, myocardial infarction within 12 months prior to the study entry, or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent. Any other concomitant serious illness or organ system dysfunction which in the opinion of the investigator would either compromise patient safety or interfere with the evaluation of the safety and anti-tumor activity of the test drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
Disease control rate after 18 weeks | 18 weeks
  To determine the disease control rate at 18 weeks of afatinib and cetuximab treatment in patients with NSCLC harboring an EGFR exon 20 insertion mutation.

SECONDARY OUTCOMES:
Objective tumor response | Scans every 6 weeks until tumor progression, start of another treatment or death.
  Objective tumor response (complete response and partial response)determined by RECIST v1.1.
Safety (intensity and incidence of adverse events) | Up to 30 days after last study drug intake.
  Safety as indicated by intensity and incidence of adverse events, graded according to NCI CTCAE Version 4.03.
Duration of response (DOR) | Scans every 6 weeks until tumor progression
  Time from documentation of tumor response to disease progression
Progression free survival | Until progression, every 6 weeks up to progression
  Time from the date of start treatment to the date of the first documented tumor progression as determined by RECIST1.1, or death due to any cause
Overall survival | Every 6 weeks up to death
  Time form date of start treatment to the date of death from any cause

OTHER OUTCOMES:
Genetic profiling to assess predictors of response and resistance - circulating free (cf)DNA | At baseline, cycle 1 day 15 and at treatment discontinuation (expected 6 months after start)
  cfDNA samples will be collected to assess predictors of response and resistance.

CONTACTS AND LOCATIONS:
Overall Officials: J de Langen, MD, PhD, Principal Investigator — NKI-AvL
Locations (4):
- Netherlands (4):
  - Antoni van Leeuwenhoek, Amsterdam, North Holland
  - VU Medical Center, Amsterdam
  - University Medical Center Groningen, Groningen
  - Maastricht UMC+, Maastricht

IPD SHARING:
Plan to Share IPD: Undecided